CLINICAL TRIAL: NCT04464239
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending and Repeated Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TS-142 Administered Orally to Healthy Male and Female Participants
Brief Title: A Single Ascending and Repeated Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TS-142 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical R&D Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TS142-US101
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Healthy Volunteers
Keywords: TS-142
MeSH Terms: interventions — TS-142

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: Cohort 1: TS-142 10 mg (Experimental): Single dose of TS-142 10 mg or placebo in a fasted condition
  Interventions: Drug: TS-142; Drug: TS-142 Placebo
- Part A: Cohort 2: TS-142 30 mg (Experimental): Single dose of TS-142 30 mg or placebo in a fasted condition.
  Interventions: Drug: TS-142; Drug: TS-142 Placebo
- Part B: Cohort 4: TS-142 20 mg (Experimental): Daily doses of 20 mg TS-142 or placebo for 7 days before bedtime.
  Interventions: Drug: TS-142; Drug: TS-142 Placebo

INTERVENTIONS:
Drug: TS-142 — TS-142 tablets
Drug: TS-142 Placebo — TS-142 matching placebo tablets

SUMMARY:
This is a study to evaluate the safety, tolerability, and pharmacokinetics of single oral doses of TS-142 compared to placebo and of a single repeated dose compared to placebo in healthy volunteers. This Phase I study is composed of two parts; Part A (Single Ascending Dose) and Part B (Repeated Dose). The study employs a randomized, double-blind, placebo-controlled, parallel group design to evaluate the single and repeat-dose safety and pharmacokinetics of TS-142 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and female participants between 18 and 55 years of age, inclusive
* Body weight ≥ 45 kg at screening and admission visits.
* Body Mass Index (BMI) ≥ 18 and ≤ 30 kg/m^2 at screening visit.

Exclusion Criteria:

* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at the screening and/or admission visits.
* Clinically significant abnormal physical examination (including neurological assessments), vital signs, or 12-lead ECGs at the screening and/or admission visits.
* QTcF >450 msec for male participants or QTcF >470 msec for female participants at the screening and/or admission visits.
* Significant history or presence of hepatic, renal, cardiovascular, pulmonary, gastrointestinal, hematological, neurological, immunologic, ophthalmologic, metabolic or oncological disease.
* History or present diagnosis of sleep disorders.
* Currently experiencing sleep disturbance related to postmenopausal symptoms at the screening and/or admission visits.
* History or presence of suicidal behavior, defined as participants who have answered 'YES' to any of the C-SSRS suicidal behavior questions at the screening and/or admission visits.
* Positive urine screen for alcohol or controlled substances at the screening or admission visits.
* Recent history (within the previous 6 months) of alcohol or drug abuse.
* Regular alcohol consumption of > 2 units/day or 10 units/week during the last 3 months prior to screening. One unit is equivalent to 8 g of alcohol: a half pint (240 mL) of beer, a glass (125 mL) of wine, or 25 mL of spirits.
* Current use, or use of tobacco or tobacco-containing products (cigarettes, pipes, e-cigarettes, nicotine patches, etc.) during the month prior to screening, or positive urine cotinine screen (>400 ng/mL) at the screening and/or admission visits.
* History of and/or current evidence of serologic positive results for hepatitis B surface antigen (HBsAg), hepatitis C antibodies, or human immunodeficiency virus (HIV) antibodies 1 and 2.
* Donation of one or more units of blood, plasma (including platelet donations), or acute loss of an equivalent amount of blood within 60 days prior to screening visit (one unit= 450 mL).
* Exposure to any investigational product within 60 days prior to screening.
* Use of any prescription or over-the-counter medication, herbal medication, vitamins, or mineral supplements within 14 days prior to administration of the study drug.
* Participants who regularly consume >500 mg of caffeine on a daily basis.
* Is known to be allergic to the study drug or any components of the study drug.
* Participated in strenuous exercise within 48 hours prior to study start (initial dosing) and/or is unwilling to avoid strenuous exercise at any time throughout the study.
* Participants who work night shifts or need to work night shifts during the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events | Part A: Day 1 to Day 10; Part B: Day 1 to Day 16
TS-142 Plasma Pharmacokinetic Profile - Cmax | Part A: Day 1 predose and at multiple time points (up to 48 hours) postdose; Part B: Day 1 predose and at multiple time points (up to 12 hours) postdose, Day 2 to Day 6 predose, Day 7 predose and at multiple time points (up to 48 hours) postdose
  Maximum plasma concentration
TS-142 Plasma Pharmacokinetic Profile - Tmax | Part A: Day 1 predose and at multiple time points (up to 48 hours) postdose; Part B: Day 1 predose and at multiple time points (up to 12 hours) postdose, Day 2 to Day 6 predose, Day 7 predose and at multiple time points (up to 48 hours) postdose
  Time to maximum plasma concentration
TS-142 Plasma Pharmacokinetic Profile - AUC(0-∞) | Part A: Day 1 predose and at multiple time points (up to 48 hours) postdose; Part B: Day 1 predose and at multiple time points (up to 12 hours) postdose, Day 2 to Day 6 predose, Day 7 predose and at multiple time points (up to 48 hours) postdose
  Area Under the Concentration vs. Time Curve from Time Zero to Infinity
TS-142 Plasma Pharmacokinetic Profile - AUC(0-last) | Part A: Day 1 predose and at multiple time points (up to 48 hours) postdose; Part B: Day 1 predose and at multiple time points (up to 12 hours) postdose, Day 2 to Day 6 predose, Day 7 predose and at multiple time points (up to 48 hours) postdose
  Area Under the Concentration vs. Time Curve from Time Zero to Last Measurable Concentration
TS-142 Plasma Pharmacokinetic Profile - AUC(0-tau) | Part A: Day 1 predose and at multiple time points (up to 48 hours) postdose; Part B: Day 1 predose and at multiple time points (up to 12 hours) postdose, Day 2 to Day 6 predose, Day 7 predose and at multiple time points (up to 48 hours) postdose
  Area Under the Concentration vs. Time Curve over a Dosing Interval
TS-142 Plasma Pharmacokinetic Profile - %AUCex | Part A: Day 1 predose and at multiple time points (up to 48 hours) postdose; Part B: Day 1 predose and at multiple time points (up to 12 hours) postdose, Day 2 to Day 6 predose, Day 7 predose and at multiple time points (up to 48 hours) postdose
  Percentage of the area extrapolated for calculation of AUC(0-∞)
TS-142 Plasma Pharmacokinetic Profile - λz | Part A: Day 1 predose and at multiple time points (up to 48 hours) postdose; Part B: Day 1 predose and at multiple time points (up to 12 hours) postdose, Day 2 to Day 6 predose, Day 7 predose and at multiple time points (up to 48 hours) postdose
  Elimination rate constant
TS-142 Plasma Pharmacokinetic Profile - t1/2 | Part A: Day 1 predose and at multiple time points (up to 48 hours) postdose; Part B: Day 1 predose and at multiple time points (up to 12 hours) postdose, Day 2 to Day 6 predose, Day 7 predose and at multiple time points (up to 48 hours) postdose
  Apparent terminal half-life
TS-142 Plasma Pharmacokinetic Profile - CL/F | Part A: Day 1 predose and at multiple time points (up to 48 hours) postdose; Part B: Day 1 predose and at multiple time points (up to 12 hours) postdose, Day 2 to Day 6 predose, Day 7 predose and at multiple time points (up to 48 hours) postdose
  Apparent oral clearance
TS-142 Plasma Pharmacokinetic Profile - Vd,z/F | Part A: Day 1 predose and at multiple time points (up to 48 hours) postdose; Part B: Day 1 predose and at multiple time points (up to 12 hours) postdose, Day 2 to Day 6 predose, Day 7 predose and at multiple time points (up to 48 hours) postdose
  Volumes of distribution
TS-142 Urine Pharmacokinetic Profile - Ae | Part A: Day 1 predose and pooled for multiple intervals (up to 48 hours) postdose
  Amount excreted in urine
TS-142 Urine Pharmacokinetic Profile - Fe% | Part A: Day 1 predose and pooled for multiple intervals (up to 48 hours) postdose
  Percent of dose excreted in urine
TS-142 Urine Pharmacokinetic Profile - CLr | Part A: Day 1 predose and pooled for multiple intervals (up to 48 hours) postdose
  Renal clearance

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Director, Study Director — Taisho Pharmaceutical R&D Inc.
Locations (1):
- PPD Phase I unit, Austin, Texas, United States